CLINICAL TRIAL: NCT05941234
Title: Improving Personalised Glioblastoma Care by Stem Cell Analysis, Omics (Including Immunomics) and Artificial Intelligence Approaches
Brief Title: Stem Cell Analysis, Omics (Including Immunomics) and Artificial Intelligence in Glioblastoma
Acronym: IPerGlioGEM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Oslo University Hospital (Other); Istituto Superiore di Sanità (Other); Luxembourg Institute of Health (Other Government); Hospital Donostia (Other); University Medical Center Goettingen (Other); National Research Council (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 5755
Record Dates: First submitted 2023-06-14; First posted 2023-07-12 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Glioblastoma, IDH-wildtype
Keywords: glioblastoma; tumor microenvironment; cancer stem cell; artificial intelligence
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients cohort Fondazione Policlinico Gemelli (Other): Collection of tumor and blood samples at T0 (surgery) and T1 (6 months follow-up) Tumor microenvironment and blood multi-omics analysis In-depth functional characterization of tumor microenvironment Cancer stem cells generation and drug testing Data integration by business intelligence and development of artificial intelligence-based prognostic markers
  Interventions: Other: Biological biomarker analysis

INTERVENTIONS:
Other: Biological biomarker analysis — Collection of tumor and blood samples at T0 (surgery) and T1 (6 months follow-up) Tumor microenvironment and blood multi-omics analysis In-depth functional characterization of tumor microenvironment Cancer stem cells generation and drug testing Data integration by business intelligence and development of AI-based prognostic markers

SUMMARY:
The study aims at:

1. Perform a multilayer analysis relying on tight integration of in-depth multi-omics approaches with clinical data to discover immune markers, with attention to age and sex differences, predicting prognosis and defining key life/environmental elements, to guide AI-driven personalised treatments and ensure improved care and QoL of glioblastoma patients.
2. To deepen glioblastoma knowledge through the study of glioblastoma stem cell cultures and to assess the sensitivity of glioblastoma stem cell cultures to a number of chemotherapeutics in different experimental conditions.
3. To create a comprehensive, stakeholder-generated guidelines for the ethical use of patient data for artificial intelligence-assisted prediction systems in glioblastoma, including an online, easily accessible patient information brochure to increase patient empowerment in the field.

ELIGIBILITY:
Inclusion Criteria:

To be enrolled in the study patients must:

1. Have a radiological diagnosis of supratentorial glioblastoma, or
2. Have a radiological diagnosis of first recurrence of a primary supratentorial glioblastoma (for which a formal histopathologic diagnosis of glioblastoma had made at first surgery), according with RANO criteria;
3. Be a candidate to neurosurgery for glioblastoma at the Operational Unit of Neurosurgery Fondazione Policlinico Gemelli IRCCS;
4. Be of an age of 18 years or above;
5. Provide written informed consent for participation to the study.

Exclusion criteria

To be enrolled in the study patients must not:

1. Have not enough pathological material removed at surgery available both for mandatory routine histopathological diagnosis and for the present study, as judged by the Principal Investigator;
2. Have not a definitive pathological diagnosis of a primary supratentorial glioblastoma, according with 2021 World Health Organization classification.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Identification of immune signatures in glioblastoma predictive of overall survival | 36 months
  Immune omic markers, namely the tumor count of the different lymphocyte subtypes and of T-cell receptor subtypes, will be correlated with overall survival.
identification of lifestyle/environmental signatures predictive of overall survival | 36 months
  A questionnaire investigating lifestyle/environmental patients features, including dietary habits, will be developed. Questionnaire data will be correlated with overall survival.
Cancer stem cell-based chemosensitivity assay | 36 months
  Assessment of the in vitro sensitivity of patient-derived cancer stem cells to chemotherapeutics

CONTACTS AND LOCATIONS:
Overall Officials: Quintino Giorgio D'Alessandris, MD, PhD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No